CLINICAL TRIAL: NCT03073616
Title: Is Lung Ultrasound the Technique of Choice for the Diagnosis of Pneumothorax Following the Nuss Procedure for Pectus Excavatum?
Brief Title: Lung Ultrasound for the Postoperative Diagnosis of Pneumothorax in Children
Acronym: ECO_NUSS
Status: Completed | Type: Observational
Sponsor: Nicola Disma, MD (Other)
Responsible Party: Sponsor-Investigator, Nicola Disma, MD, Principal Investigator, Istituto Giannina Gaslini
Organization: Istituto Giannina Gaslini (Other)
Other Study IDs: Lung-US in children
Record Dates: First submitted 2017-02-20; First posted 2017-03-08 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Pectus Excavatum
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung ultrasound: Every patient will receive a chest RX and lung US
  Interventions: Device: Lung ultrasound

INTERVENTIONS:
Device: Lung ultrasound — Lung ultrasound and chest RX

SUMMARY:
This study will be conducted to determine the advantages and limitations of sonography compared with chest radiography, in the detection of post procedure iatrogenic pneumothorax in patients underwent to Pectus Excavatum (PE) with Nuss repair.

DETAILED DESCRIPTION:
The Nuss procedure is a minimally invasive technique for the repair of Pectus Excavatum (MIRPE).

Residual pneumothorax (PNX) is reported in more than 50% after Nuss procedure. It is a consequence of the introduction of the scope and bar in the pleural space and is considered a minor complication due to the minimal clinical consequences. It is routine practice to confirm the diagnosis of PNX with a conventional chest X-Ray either in the operating room at the end of thoracic surgery or in the recovery room unit immediately after surgery.However, anterior pneumothorax can occur and chest-X ray could not be able to detected the PNX. Nowadays lung ultrasound (LUS) allows a bedside non-invasive evaluation of the patient(with a sensitivity and specificity of 92 and 99% respectively) without exposure to ionized radiation, can be performed more quickly than chest radiography and therefore can be repeated several times without additional risks. The use of LUS in pediatric age groups is more recent, but is becoming widely utilized both in neonatal and pediatric respiratory diseases.

Bedside sonography for diagnosis of PNX has been well described in emergency and trauma medicine literature and it is resulted to be more sensitive and specific than portable anteroposterior chest radiography. Although there are few studies describing the use of ultrasound for the detection of surgical pneumothorax, none of them studied its use after Nuss Procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients following Nuss procedure for PE repair at Giannina Gaslini Institute

Exclusion Criteria:

* absence of informed consent from parents
* poor quality of the pre-operatory acoustic window

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 66 consecutive pediatric patients undergoing Nuss procedure for Pectus Excavatum correction at Giannina Gaslini Institute, Genova, Italy
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Detection of PNX | 60 minutes after the end of surgery
  Detection of residual PNX immediately after surgery for NUSS repair, either using lung ultrasound (LUS): sliding (Y/N), line B (Y/N), lung pulse (Y/N), lung point (Y/N) and Rx PNX=Y/N).

SECONDARY OUTCOMES:
Lung ultrasound and operator, composite measurement | Before surgery, 60 minutes after surgery and 24 hours after surgery
  The diagnosis of "PNX" and "no PNX" has to be in agreement between operators (anesthesiologist and student)
Postoperative complications | 5 days after surgery
  Incidence of Postoperative Pulmonary Complication

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Giannina Gaslini, Genova, Italy

IPD SHARING:
Plan to Share IPD: Undecided